CLINICAL TRIAL: NCT07029919
Title: Personalized Approach To Habits - Sleep
Acronym: PATH-S
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KDH Research & Communication (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-02-02; 1R43HL174208-01 (NIH)
Record Dates: First submitted 2025-06-07; First posted 2025-06-19 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Adolescent Behavior; Sleep Disturbance; Asthma in Children; Knowledge, Attitudes, Practice; Attitude; Habits
Keywords: Teens; Adolescents; Sleep; Asthma; Habits; Support for high risk teens
MeSH Terms: conditions — Adolescent Behavior; Parasomnias; Behavior; Habits; Asthma

STUDY DESIGN:
Intervention Model Description: Teens will be randomly assigned to either the treatment group, which will be exposed to educational material on the Personalized Approach To Habits - Sleep (PATH-S app), or the control group, which will not be exposed to educational material on the PATH-S app during the study period. Both groups will complete pretest and posttest assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PATH-S Treatment (Experimental): Teens in the treatment group will be exposed to the educational material on the PATH-S app. They will engage with the app, log daily habits and sleep, and complete pretest and posttest assessments to measure changes in their knowledge, attitudes, intentions and self-efficacy.
  Interventions: Behavioral: PATH-S app
- Control (No Intervention): Teens in the control group will not be exposed to the educational material on the PATH-S app. They will engage with the app, continue their usual schedules without the additional educational material, and complete pretest and posttest assessments to measure changes in their knowledge, attitudes, intentions and self-efficacy.

INTERVENTIONS:
Behavioral: PATH-S app — PATH-S will use casual gaming and intermittent reinforcement techniques to encourage high risk teens to adopt and persist with personalized habits to improve sleep.
  Arms: PATH-S Treatment

SUMMARY:
Two arm study, intervention and control, to explore the impact of an app to help high risk teens with asthma improve their sleep

DETAILED DESCRIPTION:
The investigators will use a randomized, two-group, pretest/posttest design to test the efficacy of the Personalized Approach To Habits - Sleep (PATH-S app) and explore the following research question: To what extent does exposure to the PATH-S app increase teens' knowledge, cues to action, perceived sleepiness, and self-efficacy related to improving sleep?

PATH-S will use casual gaming and intermittent reinforcement techniques to encourage teens to adopt and persist with personalized habits to improve sleep duration. Researchers worked with subject matter experts, physicians, and the intended audience to ensure the PATH-S app reflects the specific needs of high risk teens with asthma; minimize counter-productive duplications of services and resource expenditure; and create empowered opportunities for teens to improve their overall sleep and habits.

The Principal Investigator (PI), with input from the subject matter experts and physicians, developed necessary research materials, including the recruitment protocols, evaluation instrumentation, and human subjects consent materials . The PI also outlined the appropriate statistical analysis methods. All procedure documents were reviewed by the KDH Research & Communication (KDHRC) Institutional Review Board before the evaluation launch.

Investigators will recruit participants through evaluation partners who will disseminate the study information to teens via electronic notifications and flyers. Evaluation partners include national asthma organizations. The notifications and flyers provide information about the goal of the study, participant eligibility, and a link to an eligibility form. Once a potential participant completes the eligibility form and s/he is eligible for the study, they will receive a link to a consent form located on a secure online platform.

After consent and enrollment into the study, teens will complete a pretest survey and be randomly assigned to the intervention or control group. The intervention group will be exposed to the PATH-S app, with educational material, and will complete an online posttest survey after 28 days. The control group participants will be exposed to a cloned copy of the PATH-S app, but without the educational material, and will complete an online posttest survey after 28 days. Participant responses to pretest and posttest survey measures will be linked using non-personal identifiers.

The investigators will download and export the data from Alchemer, along with data logged on the app, into encrypted Excel files and import the raw data into STATA. The investigators will match the pretest and posttest responses using the non-personal identifiers and conduct analyses to test for the effect of the PATH-S app exposure on changes in teens' knowledge, cues to action, perceived sleepiness, and self-efficacy related to improving sleep.

The initial feasibility criterion is: Statistically significant (p<0.05) and positive relationship between exposure to PATH-S app and increased knowledge among the intervention group in comparison to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Must be between 14 and 17 years old.
* Have an asthma diagnosis from a healthcare provider.
* Speak and understand English.
* Have access to a computer and the Internet.
* Have a smartphone and the ability to download and use an app.
* Live in the United States.

Exclusion Criteria:

* None

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Knowledge Pretest Score | Baseline
  Investigators will ask participants 8 multiple choice knowledge questions related to sleep health and habits which investigators will average to create a composite knowledge score for each participant ranging from 0 to 100. A score of 0 means a participant got zero questions correct while a score of 100 means a participant got all questions correct. Investigators will average these composite scores across all participants for both groups to create mean scores ranging from 0 to 100, the higher the score the more questions participants answer correctly.
Knowledge Posttest Score | Posttest- 28 days
  Investigators will ask participants 8 multiple choice knowledge questions related to sleep health and habits which investigators will average to create a composite knowledge score for each participant ranging from 0 to 100. A score of 0 means a participant got zero questions correct while a score of 100 means a participant got all questions correct. Investigators will average these composite scores across all participants for both groups to create mean scores ranging from 0 to 100, the higher the score the more questions participants answer correctly.
Cues to Action Pretest Score | Baseline
  Investigators will ask participants 9 Likert-type scale questions to measure cues to action, where they rate their level of agreement with various statements. Each answer choice rating will range from 1 to 10, with higher ratings representing higher perceptions of cues to action. Investigators will average ratings from each question to create an average composite rating for each participant ranging from 1 to 10, with 1 being the lowest score and 10 being the highest. Higher score means better outcome. Then, investigators will average these composite scores for each group.
Cues to Action Posttest Score | Posttest- 28 days
  Investigators will ask participants 9 Likert-type scale questions to measure cues to action, where they rate their level of agreement with various statements. Each answer choice rating will range from 1 to 10, with higher ratings representing higher perceptions of cues to action. Investigators will average ratings from each question to create an average composite rating for each participant ranging from 1 to 10, with 1 being the lowest score and 10 being the highest. Higher score means better outcome. Then, investigators will average these composite scores for each group.
Self-efficacy Pretest Score | Baseline
  Investigators will ask participants 6 Likert-type scale questions related to perceived self-efficacy with improving sleep health. Each rating will range from 1 to 10, with higher ratings representing higher perceptions of confidence in improving sleep health. Investigators will average ratings from each question to create an average composite rating for each participant ranging from 1 to 10, with 1 being the lowest possible score and 10 being the highest score. Higher scores mean better outcomes. Then, investigators will average these composite scores for both groups.
Self-efficacy Posttest Score | Posttest- 28 days
  Investigators will ask participants 6 Likert-type scale questions related to perceived self-efficacy with improving sleep health. Each rating will range from 1 to 10, with higher ratings representing higher perceptions of confidence in improving sleep health. Investigators will average ratings from each question to create an average composite rating for each participant ranging from 1 to 10, with 1 being the lowest possible score and 10 being the highest score. Higher scores mean better outcomes. Then, investigators will average these composite scores for both groups
Sleepiness/Restfulness Pretest Score | Baseline
  Investigators will ask participants 5 Likert-type scale questions related to perceived sleepiness or tiredness during different situations. Each rating will range from 1 to 4, with higher ratings representing higher perceptions of tiredness. Investigators will average ratings from each question to create an average composite rating for each participant ranging from 1 to 4, with 1 being the lowest possible score and 4 being the highest score. Lower scores mean better outcomes. Then, investigators will average these composite scores for both groups.
Sleepiness/Restfulness Posttest Score | Posttest- 28 days
  Investigators will ask participants 5 Likert-type scale questions related to perceived sleepiness or tiredness during different situations. Each rating will range from 1 to 4, with higher ratings representing higher perceptions of tiredness. Investigators will average ratings from each question to create an average composite rating for each participant ranging from 1 to 4, with 1 being the lowest possible score and 4 being the highest score. Lower scores mean better outcomes. Then, investigators will average these composite scores for both groups.

SECONDARY OUTCOMES:
Satisfaction at Posttest Score | Posttest- 28 days
  Investigators will ask only the intervention group participants 5 Likert-type scale questions related to their satisfaction with the PATH-S app. Each rating will range from 1 to 10, with higher scores representing higher satisfaction with the PATH-S app. Investigators will average ratings from each question to create an average composite rating for each intervention participant, then investigators will average these scores across the intervention group. Scores will range from 1 to 10, with higher scores meaning better satisfaction/outcome.

OTHER OUTCOMES:
Change in Knowledge Scores from Pretest to Posttest | Posttest- 28 days
  At both pretest and posttest, investigators will ask all participants the same 8 multiple choice knowledge questions related to sleep health and habits which investigators will average to create a composite knowledge score for each participant ranging from 0 to 100. A score of 0 means a participant got zero questions correct while a score of 100 means a participant got all questions correct. Investigators will average these composite scores across all participants for both groups to create mean scores ranging from 0 to 100, the higher the score the more questions participants answer correctly. Investigators will then subtract pretest scores from posttest scores and average these changes for all participants. Higher scores mean higher gains from baseline to posttest.
Change in Cues to Action Scores from Pretest to Posttest | Posttest- 28 days
  At both pretest and posttest, investigators will ask all participants the same 9 Likert-type scale questions to measure cues to action, where they will rate their level of agreement with various statements. Each answer choice rating will range from 1 to 10, with higher ratings representing higher perceptions of cues to action. Investigators will average ratings from each question to create an average composite rating for each participant ranging from 1 to 10, with 1 being the lowest score and 10 being the highest. Higher score means better outcome. Then, investigators will average these composite scores for each group. Investigators will then subtract pretest scores from posttest scores and average these changes for all participants. Higher scores mean higher gains from baseline to posttest.
Change in Self-Efficacy Scores From Pretest to Posttest | Posttest- 28 days
  At both pretest and posttest, investigators will ask all participants the same 6 Likert-type scale questions related to perceived self-efficacy with improving sleep health. Each rating ranged from 1 to 10, with higher ratings representing higher perceptions of confidence in improving sleep health. Investigators will average ratings from each question to create an average composite rating for each participant ranging from 1 to 10, with 1 being the lowest possible score and 10 being the highest score. Higher scores mean better outcomes. Then, investigators will average these composite scores for both groups. Investigators will then subtract pretest scores from posttest scores and average these changes for all participants. Higher scores mean higher gains from baseline to posttest.
Change in Sleepiness/Restfulness Scores From Pretest to Posttest | Posttest- 28 days
  At both pretest and posttest, investigators will ask all participants the same 5 Likert-type scale questions related to perceived sleepiness or tiredness during different situations. Each rating will range from 1 to 4, with higher ratings representing higher perceptions of tiredness. Investigators will average ratings from each question to create an average composite rating for each participant ranging from 1 to 4, with 1 being the lowest possible score and 4 being the highest score. Lower scores mean better outcomes. Then, investigators will average these composite scores for both groups. Investigators will then subtract pretest scores from posttest scores and average these changes for all participants. A positive change (i.e., a decrease in score) reflects higher gains, indicating a decrease in perceived tiredness from baseline to posttest.

CONTACTS AND LOCATIONS:
Overall Officials: Eric C. Tombly, PhD, Principal Investigator — KDH Research & Communication
Locations (1):
- KDH Research & Communication, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No